CLINICAL TRIAL: NCT00347152
Title: Overnight Versus Progressive Conversion of Multiple Daily Dose Enteric-Coated Divalproex to Once-Daily Divalproex Extended Release: Which Strategy is Better Tolerated by Patients With Intellectual Disabilities?
Brief Title: Comparison of Immediate vs Gradual Switch to Divalproex in Adults With Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Abbott (Industry)
Responsible Party: Jessica Hellings, MD, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10399
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Epilepsy
Keywords: Intellectual disabilities; development disabilities; behavior disorders; stable epilepsy
MeSH Terms: conditions — Epilepsy; Intellectual Disability; Mental Disorders | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Slow Progressive Divalproex DR to Divalproex ER switch
  Interventions: Drug: Divalproex
- 1 (Active Comparator): Immediate, Progressive Divalproex DR to Divalproex ER switch
  Interventions: Drug: Divalproex

INTERVENTIONS:
Drug: Divalproex — Divalproex, 8-20% taper
  Other Names: Depakote
  Arms: 2
Drug: Divalproex — Divalproex, 8-20% taper
  Other Names: Depakote
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether there is any difference in side effects experienced by individuals with intellectual disorders taking Depakote DR (immediate release form) when they are switched to the extended release form (ER) overnight versus when they switch more gradually over a week.

DETAILED DESCRIPTION:
Considering that there are potential advantages to once-daily depakote extended release in terms of decreased side effects, decreased medication errors and patient compliance, there is a need to determine the best method of conversion from multiple-daily dose delayed release depakote to once-daily for subjects with epilepsy bipolar disorder or behavior disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients currently taking divalproex direct release for any seizure and/or behavior disorder
* patients with intellectual disability
* other medications for co-morbid disease are permitted, provided no plans for changes in medication used for the treatment of the disorder are expected

Exclusion Criteria:

* patients with a recent history of status epilepticus in the past 6 months
* seizures in the past 3 months
* patients with acute illness requiring changes in concurrent drugs
* patients unwilling to change from their present direct release divalproex to divalproex extended release
* patients that do not have a reliable caregiver
* patients with lack of verbal expressive speech

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
direct observation of side effects by staff and investigator, side effect ratings using the MOSES side effect rating scale post-switch. (Multidimensional observational scale for elderly subjects) | Baseline to day +8

SECONDARY OUTCOMES:
seizures observed, compared with prior rate of seizures;maintenance of clinical response using the Clinical Global Impressions Scale-improvement subscale; | Baseline to day + 8
total valproic acid serum levels (trough of pre-dose measurements) | Prior to conversion, 1 week post conversion
changes in blood work, including CBC, platelet counts, LFT, serum chemistry panel | Prior to and one week post conversion

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Hellings, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States